CLINICAL TRIAL: NCT07282171
Title: An Open-Label, Dose Finding Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Ascending Subcutaneous Doses of CBP-4888 in Hospitalized Participants With Preterm Preeclampsia Receiving Standard of Care, Expectant Management
Brief Title: A Study to Investigate the Safety, Pharmacodynamic and Pharmacokinetic Characteristics of CBP-4888 in Hospitalized Participants With Preterm Preeclampsia and Their Children up to 24 Months
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Comanche Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBP-4888-101
Record Dates: First submitted 2025-11-17; First posted 2025-12-15 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: sFlt1 Mediated Preterm Preeclampsia; Preeclampsia; Preterm Preeclampsia
Keywords: preterm preeclampsia; Hypertensive disorder of pregnancy; Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia; Toxemia

STUDY DESIGN:
Intervention Model Description: The study will follow a single ascending dose design, with up to 60 participants enrolled across 6 dose levels. For each of the planned dose levels, all 4 participants will receive a subcutaneous dose of IP (CBP-4888) + standard of care (SOC)/Expectant Management + additional safety surveillance.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CBP-4888 (Experimental): On Day 1, participants will receive a subcutaneous dose of CBP-4888.
  Interventions: Drug: CBP-4888

INTERVENTIONS:
Drug: CBP-4888 — Participants will receive a subcutaneous dose of CBP-4888. Dosing is weight based using the participant's first trimester weight.

SUMMARY:
This study is a dose finding study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of subcutaneous CBP-4888 in hospitalized participants with Preterm Preeclampsia receiving Standard of Care, Expectant Management. Eligible participants are between 26 +0/7 and 35 +6/7 weeks gestational age and clinically appropriate for inpatient expectant management. Eligible participants will receive standard of care expectant management for their pregnancy with the only study interventions being one subcutaneous dose of CBP-4888.

Participants will:

* receive a single subcutaneous injection dose of CBP-4888 and will be followed through delivery and for 42 days (+14 days) after delivery. Participants will be followed through 6 weeks post delivery.
* Infants will be evaluated immediately postpartum and then followed through 24 months of age with standard infant and pediatric assessments with phone calls made to parents.

DETAILED DESCRIPTION:
An Open-Label, Dose Finding Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Subcutaneous CBP-4888 in Hospitalized Participants with Preterm Preeclampsia Receiving Standard of Care, Expectant Management. The study will follow a single ascending dose design, with up to 60 participants enrolled across 6 dose level groups. For each of the planned six dose levels, all 4 participants will receive a single SC injection dose of IP (CBP-4888) + standard of care (SOC)/Expectant Management + additional safety surveillance for the mother and neonate through delivery and for 42 days (+14 days) after delivery. Infants will be followed for up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized with a hypertensive disorder of pregnancy (preeclampsia) defined by elevated blood pressure after 20 weeks gestation with proteinuria or, in the absence of proteinuria, with evidence of organ dysfunction (e.g., thrombocytopenia, renal insufficiency, or impaired liver function), and expected to remain hospitalized through delivery
* The subject has given written consent to participate in the study.
* Pregnant participants aged 18 to 45 years of age
* Gestational age at Day 1 between 26 weeks 0/7 days and 35 weeks 6/7 days
* Deemed clinically stable and suitable for expectant management for at least 72 hours post CBP-4888 administration
* The woman carries a singleton pregnancy
* Anticipate that hospitalization will continue through delivery

Exclusion Criteria:

* Placenta previa, abruption, accreta, or persistent unexplained vaginal bleeding.
* Fetal growth restriction (<3rd percentile, or <10th percentile with abnormal Doppler) or known major chromosomal/genetic abnormalities.
* Maternal conditions requiring immediate delivery (e.g., severe hypertension, eclampsia, non-reassuring fetal status, pulmonary edema).
* Known active maternal infections considered to potentially affect placental function.
* Significant maternal medical conditions (e.g., HELLP syndrome, advanced kidney disease, severe cardiac disease, uncontrolled neurological disorder, lupus with nephritis/cerebritis).
* Use of another investigational drug within 30 days prior to study entry.
* Any other condition that, in the investigator's judgment, poses risk to mother or fetus.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment emergent events and adverse events of special interest when CBP-4888 is administered to pregnant participants | 6 weeks postpartum
  Incidence of treatment-emergent adverse events (TEAEs) in pregnant participants receiving subcutaneous CBP-4888 through delivery (up to 6 weeks postpartum).
Determine recommended phase 2 dose | From pre-dose on Day 1 through the last measurable concentration at approximately 72 hours postpartum in serum
  To characterize the pharmacodynamic effect of CBP-4888 on maternal plasma sFlt1 levels

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) of siRNA-2283 siRNA-2519 | From pre-dose on Day 1 through the last measurable concentration at approximately 120 hours post-dose
  To characterize the PK in plasma of CBP-4888
Incidence of Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESIs) in Infants Exposed In Utero to CBP-4888 | From birth through 180 days of age
  Infants born to participants who received CBP-4888 during pregnancy will be assessed for SAEs and AESIs to investigate long term safety of children of pregnant participants who were administered CBP-4888
Time to Peak Concentration (Tmax) of siRNA-2283 siRNA-2519 | From pre-dose on Day 1 through the last measurable concentration at approximately 120 hours post-dose
  To characterize PK in plasma of CBP-4888
Area Under the Concentration (AUC)-Time Curve to Last Measurable Concentration of siRNA-2283 and siRNA-2519 | From pre-dose on Day 1 through the last measurable concentration at approximately 120 hours post-dose
  To Characterize PK in plasma of CBP-4888
Neurodevelopmental Outcomes Assessed by the Ages and Stages Questionnaire (ASQ-3) to investigate long term safety of children of pregnant participants who were administered CBP-4888 | From birth through 24 months of age
  Neurodevelopment will be evaluated using the Ages and Stages Questionnaire, (ASQ-3), a validated parent-completed developmental screening tool.

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - The Royal Women's Hospital, Parkville, Victoria
  - Royal Melbourne, Melbourne

IPD SHARING:
Plan to Share IPD: Undecided